CLINICAL TRIAL: NCT06966284
Title: A Retrospective, Observational, Post-Marketing Study to Assess the Efficacy and Safety of Intravenous Infusions Polymyxin B and Colistin Methanesulfonate in Patients With Carbapenem-Resistant Gram-Negative Bacterial Infection
Brief Title: A Post-Marketing Study to Assess the Efficacy and Safety of Intravenous Polymyxin B and Colistin Methanesulfonate in Patients With Carbapenem-Resistant Gram-Negative Bacterial Infection
Status: Not yet recruiting | Type: Observational
Sponsor: TTY Biopharm (Industry)
Responsible Party: Sponsor
Other Study IDs: TTYPX2203
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Bacteremia Caused by Gram-Negative Bacteria; Bacterial Pneumonia
Keywords: polymyxin B sulfate
MeSH Terms: conditions — Pneumonia, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experiment: Polymyxin B
- Comparator: colistin methanesulfonate

SUMMARY:
This is a retrospective, observational, post-marketing study to evaluate the clinical response, microbiological response, mortality, and safety of intravenous polymyxin B and colistin methanesulfonate in patients with carbapenem-resistant gram-negative bacterial infection. Subgroup analysis by sites of infection, infectious pathogens, and baseline renal function will also be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 18 years of age.
2. Patient diagnosed with bacterial pneumonia and/or bacteremia, or other physician judged serious infection (except urinary tract infection, UTI) caused by Carbapenem-Resistant Gram-Negative Bacteria (CR-GNB).

   CR-GNB: Resistant to at least one of the carbapenem antibiotics or produce a carbapenemase (an enzyme that can make them resistant to carbapenem antibiotics).

   Diagnosis Criteria of HABP/VABP:

   • Met the clinical diagnosis criteria for HABP/VABP. HABP: Acute bacterial pneumonia in a subject hospitalized for more than 48 hours or developing within 7 days after discharge from a hospital. Subject could have experienced acute respiratory failure and required mechanical ventilation for HABP.

   VABP: Acute bacterial pneumonia in a subject receiving mechanical ventilation via an endotracheal (or nasotracheal) tube for a minimum of 48 hours.
   * ≥ 1 of the following clinical features: new onset or worsening of pulmonary symptoms or signs, hypoxemia, need for acute changes in the ventilator support system to enhance oxygenation, new onset of or increase in suctioned respiratory secretions.
   * ≥ 1 of the following signs: documented fever, hypothermia, WBC ≥ 10,000 cells/mm3, WBC ≤ 4500 cells/mm3, >15% immature neutrophils(bands)
   * CXR or lung CT: presence of new or progressive infiltrates suggestive of bacterial pneumonia.

   Diagnosis Criteria of BSI/Bacteremia: the BSI/sepsis category included bacteremia or sepsis caused by infections other than HABP/VABP, or UTI:
   * Documented BSI caused by a carbapenem-resistant Gram-negative pathogen; or
   * Systemic response to infection, meeting the clinical criteria of SIRS and an identified infection source (eg, severe skin infection, intra-abdominal infection) caused by a carbapenem-resistant Gram-negative pathogen.
3. Patient received intravenous polymyxin B or CMS treatment for ≥72 h.
4. Administration of polymyxin B or CMS within 7 days from the infection onset day.

Infection onset day: The date of specimen collection for index pathogen.

Exclusion Criteria:

1. Patient with bacteremia caused by urinary tract infection.
2. CR-GNB known to be resistant to polymyxin B or CMS.
3. Patient has infectious disease (s) caused by the following gram-negative bacteria which are known to have no response to polymyxin B and/or colistin treatment: Proteus spp., Providencia spp., Morganella spp., Serratia marcescens, Burkholderia spp., and Neisseria spp.
4. Intravenous administration of polymyxin B or colistin more than 28 days.
5. Both the treatment efficacy and safety could not be evaluated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Intent-To-Treat (ITT) population
  2. Total enrolled population
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate of polymyxin B and CMS treatment groups at TOC | TOC: End of Treatment + 7 days
Microbiological response rate of polymyxin B and CMS treatment groups at TOC | TOC: End of Treatment + 7 days
All-cause mortality of of polymyxin B and CMS treatment groups at Day 28 | Day 28 from start of treatment
Clinical response rate of polymyxin B group by sites of infection and infectious pathogens at TOC | End of Treatment + 7 days
Microbiological response rate of polymyxin B group by sites of infection and infectious pathogens at TOC | End of Treatment + 7 days
Infection-related mortality of two treatment groups at Day 28 | Day 28 from start of treatment

SECONDARY OUTCOMES:
Clinical response rate (Day 7, Day 14, Day 28, and EOT) of two treatment groups | Day 7, Day 14, Day 28, and EOT
Clinical response rate (Day 7, Day 14, Day 28 and EOT) of polymyxin B group by sites of infection and infectious pathogens | Day 7, Day 14, Day 28, and EOT
Clinical response rate (Day 7, Day 14, Day 28, EOT, and TOC) of polymyxin B group by baseline renal function | Day 7, Day 14, Day 28, EOT, and TOC
Microbiological response rate (Day 7, Day 14, and EOT) of two treatment groups | Day 7, Day 14, and EOT
Microbiological response rate (Day 7, Day 14, and EOT) of polymyxin B group by sites of infection and infectious pathogens | Day 7, Day 14, and EOT
Microbiological response rate (Day 7, Day 14, EOT, and TOC) of polymyxin B group by baseline renal function | Day 7, Day 14, EOT, and TOC
All-cause mortality (Day 14) of two treatment groups | Day 14 from start of treatment
All-cause mortality (Day 14, Day 28) of polymyxin B group by sites of infection, infectious pathogens, and baseline renal function | Day 14, Day 28 from start of treatment
Infection-related mortality (Day 14) of two treatment groups | Day 14 from start of treatment
Infection-related mortality (Day 14, Day 28) of polymyxin B group by sites of infection, infectious pathogens, and baseline renal function | Day 14, Day 28 from start of treatment